

General Consent Form Template Version Date: January 2019

Protocol Title: Assessment and Augmentation of Lip Appearance in Specific

Study Populations

Principal Investigator: Dieter Manstein, MD, PhD

Site Principal Investigator: N/A

Description of Subject Population: Healthy Volunteers

### NCT04839692

### **About this consent form**

Please read this form carefully. It tells you important information about a research study. A member of our research team will also talk to you about taking part in this research study. People who agree to take part in research studies are called "subjects." This term will be used throughout this consent form.

Partners HealthCare System is made up of Partners hospitals, health care providers, and researchers. In the rest of this consent form, we refer to the Partners system simply as "Partners."

If you decide to take part in this research study, you must sign this form to show that you want to take part. We will give you a signed copy of this form to keep.




## **Key Information**

Taking part in this research study is up to you. You can decide not to take part. If you decide to take part now, you can change your mind and drop out later. Your decision won't change the medical care you get within Partners now or in the future.

The following key information is to help you decide whether or not to take part in this research study. We have included more details about the research in the Detailed Information section that follows the key information.

### Why is this research study being done?

In this research study we want to learn more about the effects of aging and lip filler treatment on lips and the surrounding skin by comparing, among two different age groups of people, changes in the blood vessels and nerves, volume, color and texture change before and after lip filler treatment and pain tolerance from lip filler treatment. Also, we want to evaluate how oxytocin (a hormone) levels change during and after an aesthetic procedure and patient satisfaction after the procedure.

We are asking you to take part in this research study as a healthy volunteer because we need to assess healthy lips and surrounding skin across these two different groups of people in order to understand how healthy lips and surrounding skin varies across age ranges. Up to 60 people will take part in this study.

## How long will you take part in this research study?

If you decide to join this research study, it will take you about 2 weeks to complete the study. During this time, we will ask you to make 2 in-person study visits to MGH's Clinical Unit for Research Trials & Outcomes in Skin (CURTIS) at 50 Staniford Street, Suite 240 Boston, MA 02114 OR Translational Clinical Research Center (TCRC) on the 12th floor of the White Building. The first visit will take about 1 hour 30 minutes. The second visit will be scheduled for about 2 weeks after the first visit and will take up to 1 hour. There will be one follow-up call 3-7 days after visit 1 that will last about 30 minutes. Study visits will require up to 3 hours total of your time.




### What will happen if you take part in this research study?

If you decide to join this research study, the following things will happen:

- Ask you about your medical history, demographics and medications
- Review inclusion/exclusion criteria
- Non-invasive imaging of your blood vessels (OCT Imaging) of the lips and surrounding area
- Non-invasive three-dimensional imaging of the lips and surrounding area using the Cherry Imaging system
- Digital photography of lips and surrounding area
- Placement of venous access (IV placement) 4 samples of blood will be collected
- Hyaluronic Acid Lip Filler (Restylane Kysse)
- Lip volume assessment
- Pain tolerance recorded
- Patient satisfaction and self-reported color change record

### Why might you choose to take part in this study?

We cannot promise any benefits to you from taking part in this research study. However, possible benefits may include improved appearance of the lips. Others getting lip filler treatments for lip aging may benefit in the future from what we learn in this study.

## Why might you choose NOT to take part in this study?

Taking part in this research study has some risks and requirements that you should consider carefully.

Important risks and possible discomforts to know about include pain during procedure (or during IV placement), redness, swelling, lumps/bumps, bruising, itching, allergic reaction, or discoloration.

A detailed description of side effects, risks, and possible discomforts can be found later in this consent form in the section called "What are the risks and possible discomforts from being in this research study?"

Other things to consider are that study visits will require up to 3 hours total of your time.

## What other treatments or procedures are available for your condition?

We are looking for healthy volunteers and we are not treating a medical condition.




# If you have questions or concerns about this research study, whom can you call?

You can call us with your questions or concerns. Our telephone numbers are listed below. Ask questions as often as you want.

Dieter Manstein, MD, PhD is the person in charge of this research study. You can call him at (617)726-4893 on Monday through Friday 9am – 5pm. You can also call Neera Nathan, MD, MSHS at (617) 726-4454 on Monday through Friday 9am – 5pm with questions about this research study.

If you have questions about the scheduling of appointments or study visits, call Lais Gomes at (617) 726-4454.

If you want to speak with someone **not** directly involved in this research study, please contact the Partners Human Research Committee office. You can call them at 857-282-1900.

You can talk to them about:

- Your rights as a research subject
- Your concerns about the research
- A complaint about the research
- Any pressure to take part in, or to continue in the research study

Subject Identification


### **Detailed Information**

A description of this clinical trial will be available on *http://www.ClinicalTrials.gov*, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

### Why is this research study being done?

We are doing this research study to examine the effects of aging on the lips and surrounding area. In addition to examining the effects of lip filler treatment on the appearance of aging lips and pain tolerability of the treatment. We want to compare changes in lip color, texture and volume before and after filler with non-invasive imaging, including digital photography, OCT imaging and three-dimensional imaging. Also, we want to evaluate how oxytocin levels change during and after an aesthetic procedure and patient satisfaction after the procedure.

The hyaluronic acid lip filler (Restylane Kysse) is approved by the U.S. Food and Drug Administration (FDA) for lip augmentation or fuller lips. The non-invasive OCT imaging device used to take pictures of your blood vessels is not approved by the FDA for use in people but has been used previously for research on more than 1000 people.

## Who will take part in this research?

We are asking you to take part in this research study as a healthy volunteer who is eligible for lip filler treatment using the Restylane Kysse lip filler applied to the lips and surrounding skin. Up to 60 subjects will participate in this study. The study will be funded by discretionary lab funds and will not use industry funds or grant funds.

### What will happen in this research study?

### **Screening Visit (video/phone call)**

During the screening visit, the investigator will discuss the nature of the study, its requirements and its restrictions. The following will be discussed to determine if you qualify for the study:

- Review of inclusion/exclusion criteria with you
- Ask you about your medical history, medications and demographics
- Examine your lips and lip volume

After the screening, if you qualify and are interested in participating in the study we will give you consent forms to fill out and schedule visit 1. If you don't qualify, the study doctor will tell you why.




#### Visit 1

Visit 1 will take up to 1 hour 30 minutes. At this visit, we will:

- Review your medical history, medications and demographics, and the inclusion/exclusion criteria with you
- Photograph the blood vessels of your lips and surrounding area with OCT Imaging device
- Photograph your lips and surrounding area with a three-dimensional camera (Cherry Imaging system) before and right after the lip filler treatment
- Photograph your lips and surrounding area with a camera
- Placement of venous access 4 samples of blood will be collected to analyze serum oxytocin levels: before the procedure, immediately after the filler procedure,5 min and 30 min after the procedure.
- Perform hyaluronic acid lip filler (Restylane Kysse) treatment on your lips and surrounding area
- Lip volume assessment
- Ask you about the level of pain you feel with the first insertion of the filler and the overall treatment
- Record 15-30 seconds-video from your face and lips after the lip filler procedure. The video recording is optional.
- Give you aftercare instructions, stipend and parking voucher if needed
- Schedule your second visit to take place about 2 weeks after the first study visit

### Follow-up Call (3-7 days after visit 1)

The follow-up call will take up to 30 minutes. At this visit, we will ask you if you are experiencing any post-treatment pain or side effects. If you are experiencing any negative side effects we will evaluate and treat you by following standard medical procedures.

### Visit 2 (2 weeks after visit 1)

Visit 2 will take up to 1 hour. At this visit, we will:

- Photograph the blood vessels of your lips and surrounding area with OCT Imaging device
- Photograph your lips and surrounding area with a three-dimensional camera (Cherry Imaging system)
- Photograph your lips and surrounding area with a camera
- Lip volume assessment
- Ask you some questions related to your satisfaction with the procedure

Partners has an electronic system that lets your study doctors know if you are admitted to a Partners Hospital, or if you visit a Partners Hospital Emergency Department. We want to make

<sup>\*</sup>Subjects who fulfill all inclusion and exclusion criteria may enroll and begin the Visit 1 procedures that same day.




sure the study doctors know about any possible problems or side effects you experience while you are taking part in the study.

### Study Information Included in Your Electronic Medical Record

A notation that you are taking part in this research study may be made in your electronic medical record. Information from the research that relates to your general medical care may be included in the record (for example: list of allergies, results of standard blood tests done at the hospital labs).

## How may we use and share your samples and health information for other research?

The information we collect in this study may help advance other research. If you join this study, we may remove all information that identifies you (for example, your name, medical record number, and date of birth) and use these de-identified samples and data in other research. It won't be possible to link the information or samples back to you. Information and/or samples may be shared with investigators at our hospitals, at other academic institutions or at for-profit, commercial entities. You will not be asked to provide additional informed consent for these uses.

## Will you get the results of this research study?

No. The research study we are doing is only a stepping stone in understanding the lip aging process. Therefore, no information about the results of this research study or the results of your individual participation in the research study will be given to you or your doctor. Tests done for the research using your samples will not be useful in directing your medical treatment. The results of the tests will not be placed in your medical record.

# What are the risks and possible discomforts from being in this research study?

### **Lip Filler Treatment**

You will experience sharp pain and mild pressure from the first injection, which will go away with the following injections as the numbing takes effect with the anesthetic in the filler. You should immediately inform us if you experience unbearable pain or discomfort during the treatment.

Please refer to the frequency categories listed below for reporting of possible side effects/risks:




- a. Very Common (more than 1 out of 10 people)
- b. Common (between 1 and 10 out of 100 people)
- c. Uncommon (between 1 and 10 out of 1,000 people)
- d. Rare but Serious (less than 1 out of 1,000 people)

Possible side effects/risks of Restylane Kysse lip filler include:

- Very Common (more than 1 out of 10 people)
  - o Redness, pain/tenderness,
  - o Swelling,
  - o Lumps/bumps, bruising, itching, or discoloration,
  - o Change in skin tone (i.e. erythema).
- Rare but serious (less than 1 out of 1,000 people)
  - Allergic reaction\*,
  - o Infection,
  - o Scarring,
  - o Skin ulceration,
  - o Ischemia,
  - o Infarction,
  - Localized skin necrosis.

Lip fillers in the lips and perioral area are considered to be low risk but rare instances of localized skin necrosis are possible. In this case, if there are symptoms of occlusions, intense pain, or purple patches upon injection, we will have hyaluronidase (FDA approved for vascular occlusion necrosis) available in clinic to treat you.

### IV placement

The IV access can cause pain during its placement. Possible risk may include infections, bleeding and thrombophlebitis but they are rare in healthy patients. Adverse outcomes will be treated according to standard medical care.

### **OCT Imaging**

You may experience some discomfort from the pressure applied to the lips to take photographs of the blood vessels. No harm will be caused from the pressure applied. Possible risk may include allergic reaction\* to glycerol or Tegaderm (transparent film dressing) used during this imaging procedure.

### **Cherry Imaging**

There are no known risks of the three-dimensional imaging system (Cherry imaging) other than psychological distress from seeing a high-resolution photo that may highlight imperfections.




#### Non-Medical

There is a potential risk of loss of privacy. We will protect your privacy by labeling samples, information, and data files only with a study subject number code, and keeping the key to the code in a password protected database.

\*If there are any allergic reactions, we will treat you with standard medical procedures.

## What are the possible benefits from being in this research study?

We cannot promise any medical benefits to you from taking part in this research study. However, possible benefits may include improved appearance of the lips. This study can benefit future studies in the process of understanding and improving the condition of aging lips and surrounding skin, and/or reverse certain aging processes we can detect in the skin. This study may also help in understanding pain tolerance with the lip filler treatment to improve pain management techniques in the future as needed.

# Can you still get medical care within Partners if you don't take part in this research study, or if you stop taking part?

Yes. Your decision won't change the medical care you get within Partners now or in the future. There will be no penalty, and you won't lose any benefits you receive now or have a right to receive.

We will tell you if we learn new information that could make you change your mind about taking part in this research study.

## What should you do if you want to stop taking part in the study?

If you take part in this research study, and want to drop out, you should tell us. We will make sure that you stop the study safely. We will also talk to you about follow-up care, if needed.

Also, it is possible that we will have to ask you to drop out of the study before you finish it. If this happens, we will tell you why. We will also help arrange other care for you, if needed.

## Will you be paid to take part in this research study?



General Template Version Date: December 2008

You will be paid \$50 for completing all imaging activities and filler treatment during visit 1, and \$100 for completing visit 2. This means we will pay you \$150 if you complete the study visits 1 through 2. We will also provide a parking voucher for MGH main campus for each visit upon request.

We may be using an approved, outside vendor (Forte Research) to make these payments to you via a reloadable credit card-based system, called Forte Payments. This secure system is similar to a gift card or credit card.

If you are paid by this system, you will be given a Forte Payments Visa card (which is just like a debit card) when you enroll in the study. Once the card is activated, the study team will add a payment after each paid visit you complete. The payment should be available to you within one (1) business day. Research staff will not know where you spend the money. You may use the card anywhere Visa cards are accepted, such as at a grocery store. If your card is lost or stolen, please call (617) 726-4454.

We will need to collect your Social Security number in order to make these payments, and it will be shared securely with the company that runs the card-based system. Payments like this are considered taxable income. If you receive more than \$600, the payment will be reported to the IRS as income by the hospital.

We may use your samples and information to develop a new product or medical test to be sold. The Sponsor, hospital, and researchers may benefit if this happens. There are no plans to pay you if your samples or information are used for this purpose.

### What will you have to pay for if you take part in this research study?

Study funds will pay for certain study-related items and services. We may bill your health insurer for, among other things, routine items and services you would have received even if you did not take part in the research. You will be responsible for payment of any deductibles and copayments required by your insurer for this routine care or other billed care. If you have any questions about costs to you that may result from taking part in the research, please speak with the study doctors and study staff. If necessary, we will arrange for you to speak with someone in Patient Financial Services about these costs.

What happens if you are injured as a result of taking part in this research study?




We will offer you the care needed to treat any injury that directly results from taking part in this research study. We reserve the right to bill your insurance company or other third parties, if appropriate, for the care you get for the injury. We will try to have these costs paid for, but you may be responsible for some of them. For example, if the care is billed to your insurer, you will be responsible for payment of any deductibles and co-payments required by your insurer.

Injuries sometimes happen in research even when no one is at fault. There are no plans to pay you or give you other compensation for an injury, should one occur. However, you are not giving up any of your legal rights by signing this form.

If you think you have been injured or have experienced a medical problem as a result of taking part in this research study, tell the person in charge of this study as soon as possible. The researcher's name and phone number are listed in the beginning of this consent form.

### If you take part in this research study, how will we protect your privacy?

Federal law requires Partners to protect the privacy of health information and related information that identifies you. We refer to this information as "identifiable information."

### In this study, we may collect identifiable information about you from:

- Past, present, and future medical records
- Research procedures, including research office visits, tests, interviews, and questionnaires

## Who may see, use, and share your identifiable information and why they may need to do so:

- Partners researchers and staff involved in this study
- The sponsor(s) of the study, and people or groups it hires to help perform this research or to audit the research
- Other researchers and medical centers that are part of this study
- The Partners ethics board or an ethics board outside Partners that oversees the research
- A group that oversees the data (study information) and safety of this study
- Non-research staff within Partners who need identifiable information to do their jobs, such as for treatment, payment (billing), or hospital operations (such as assessing the quality of care or research)




- People or groups that we hire to do certain work for us, such as data storage companies, accreditors, insurers, and lawyers
- Federal agencies (such as the U.S. Department of Health and Human Services (DHHS) and agencies within DHHS like the Food and Drug Administration, the National Institutes of Health, and the Office for Human Research Protections), state agencies, and foreign government bodies that oversee, evaluate, and audit research, which may include inspection of your records
- Public health and safety authorities, if we learn information that could mean harm to you or others (such as to make required reports about communicable diseases or about child or elder abuse)
- Other:

Some people or groups who get your identifiable information might not have to follow the same privacy rules that we follow and might use or share your identifiable information without your permission in ways that are not described in this form. For example, we understand that the sponsor of this study may use your identifiable information to perform additional research on various products or conditions, to obtain regulatory approval of its products, to propose new products, and to oversee and improve its products' performance. We share your identifiable information only when we must, and we ask anyone who receives it from us to take measures to protect your privacy. The sponsor has agreed that it will not contact you without your permission and will not use or share your identifiable information for any mailing or marketing list. However, once your identifiable information is shared outside Partners, we cannot control all the ways that others use or share it and cannot promise that it will remain private.

Because research is an ongoing process, we cannot give you an exact date when we will either destroy or stop using or sharing your identifiable information. Your permission to use and share your identifiable information does not expire.

The results of this research study may be published in a medical book or journal, or used to teach others. However, your name or other identifiable information **will not** be used for these purposes without your specific permission.

### **Your Privacy Rights**

You have the right **not** to sign this form that allows us to use and share your identifiable information for research; however, if you don't sign it, you can't take part in this research study.

## **Partners HealthCare System Research Consent Form** Subject Identification **General Consent Form Template Version Date: January 2019** You have the right to withdraw your permission for us to use or share your identifiable information for this research study. If you want to withdraw your permission, you must notify the person in charge of this research study in writing. Once permission is withdrawn, you cannot continue to take part in the study. If you withdraw your permission, we will not be able to take back information that has already been used or shared with others, and such information may continue to be used for certain purposes, such as to comply with the law or maintain the reliability of the study. You have the right to see and get a copy of your identifiable information that is used or shared for treatment or for payment. To ask for this information, please contact the person in charge of this research study. You may only get such information after the research is finished. **Informed Consent and Authorization Statement of Person Giving Informed Consent and Authorization** • I have read this consent form. • This research study has been explained to me, including risks and possible benefits (if any), other possible treatments or procedures, and other important things about the study. • I have had the opportunity to ask questions. • I understand the information given to me.

## **Signature of Subject:**

I give my consent to take part in this research study and agree to allow my health information to be used and shared as described above.

Subject

Date

Time (optional)

| Partners HealthCare System<br>Research Consent Form | | |
|---|---|---|
| General Template<br>Version Date: December 2008 | | Subject Identification |
| Signature of Study Doctor: | | |
| Statement of Study Doctor Obtaining Consent | | |
| <ul> <li>I have explained the research to the study s</li> <li>I have answered all questions about this res</li> </ul> | • | o the best of my ability. |
| Study Doctor Obtaining Consent | Date | Time (optional) |
| Optional Video Recording Procedure Co The video recording procedure is optional and you not to have the video recording (after you lip filler below. I am interested in participating in the video recordi to take part the video recording. | can still part<br>procedure ha | s been completed). Please initial |
| Initial Date | | |
| <u>OR</u> | | |
| I am NOT interested in participating in the video rein the video recording procedure. | ecording. I ar | n initialing below to not take part |
| Initial Date | | |

### Video Recording Release:

In addition to using my video recording for this study (for study staff analysis), I give my consent for the use of my video recording for the following purposes:

| Identificat |
|-------------|


- medical or pharmaceutical publications, or presentations in conferences O YES O NO
- Educating health care professionals (such as physicians and nurses) through electronic materials (iPads), brochures and the healthcare professional website OYES O NO

Date/Time

 Patient-focused websites and patient-handouts / industry ads O YES ONO

I understand that I will not be entitled to receive any payment for the use of my video recording.

Consent Form Version:

3

Subject

Consent Form Version Date:

January 18, 2022